CLINICAL TRIAL: NCT06613256
Title: Characterisation of Endothelial Cells in Different Inflammatory Pathologies
Acronym: JEDI-2
Status: Recruiting | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 24SURN320251
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; Vasoplegia
MeSH Terms: conditions — Sepsis; Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. RNA extracted from endothelial cell biopsies
  2. Serum and plasma from paired blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Part 1 - control patients: 25 healthy volunteers
  1 X Endothelial cell biopsy
  Interventions: Other: Endothelial cell biopsy
- Part 1 - surgical patients: 20 surgical patients
  1 X Endothelial cell biopsy
  Samples collected at 24 hours post knife to skin to capture peak inflammation
  Interventions: Other: Endothelial cell biopsy
- Part 1 - sepsis patients: 20 sepsis patients
  1 X Endothelial cell biopsy
  Samples collected on admission to ICU
  Interventions: Other: Endothelial cell biopsy
- Part 2 - surgical patients: 20 surgical patients 3 X Endothelial cell biopsy
  Samples collected pre-surgery, 24 hours and 48 hours post knife to skin
  Interventions: Other: Endothelial cell biopsy
- Part 2 - sepsis patients: 20 sepsis patients 3 X Endothelial cell biopsy
  Samples collected on admission, 24 hours and 48 hours post admission to ICU
  Interventions: Other: Endothelial cell biopsy

INTERVENTIONS:
Other: Endothelial cell biopsy — Endothelial cell sample collected from the antecubital fossa of patients. A vein in the antecubital fossa is cannulated with a 20 g valveless cannula. A metal guidewire is then passed into the vessel to collect endothelial cells for analysis

SUMMARY:
The goal of this observational study is to characterise changes in gene expression in endothelial cells in patients with either sepsis or post major abdominal surgery.

The main question we plan to answer is: 'What molecular pathways are differentially expressed during inflammatory pathologies?'

DETAILED DESCRIPTION:
The immune system is a complex network of cells and molecules that protects the body from infection and injury. When the immune system is activated, it produces inflammation, which is a natural response to help heal the body. However, too much inflammation can be harmful and lead to serious complications, such as sepsis, low blood pressure, organ failure and death.

The interaction of cells that line the blood vessels (endothelial cells, EC) with the immune system, is believed to be the root cause of these symptoms. When exposed to inflammation, the instructional molecules (RNA) inside the EC change. This leads to a change of operation promoting the severe symptoms previously mentioned.

Researchers have developed new safe techniques to collect these cells from the blood vessels of patients to study disorders like diabetes, heart disease and stroke. This technique involves gently inserting a metal guidewire into an arm vein to collect ECs.

This study plans to collect ECs from patients undergoing surgery or admitted to intensive care. We also plan to collect control samples from healthy volunteers. Samples will be collected over the duration of the patients to RSFT. The RNA will be removed from the cells and counted to highlight changes in instructions in the cells.

Data from this study will potentially highlight new pathways involved in inflammation and help classify how some patients will react to current treatments. To obtain this data, this study will be split into 2 parts. Part 1 focuses on collecting one sample from a patient when they are at their most unwell states and comparing that to a sample from a healthy person. Part 2 will focus on key mRNA molecules identified during Part 1 and identifying how their expression changes over time.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteer

* Adult ≥ 18 years
* Able and willing to give consent

Surgical patients

* Adult ≥ 18 years
* Patients admitted to RSFT for planned major surgery

Critically ill patients

* Adult ≥ 18 years
* Emergency admission to ICU at RSFT
* Meets the sepsis 3.0 definition

Exclusion Criteria:

Healthy volunteer

* Not currently a patient within the hospital
* Absence of inflammatory diseases and disorders including but not limited to arthritis, peripheral artery disease, vasculitis, diabetes, cardiovascular disease and CKD.
* Not on immunomodulatory medications, such as corticosteroids
* History of recent major trauma within the last 2 months (e.g., surgery or injury requiring hospitalisation)

Surgical patients

* Patients with restricted liberty, prisoners or under legal protection
* Anticipated prohibitively difficult venous cannulation
* Presenting with inflammatory diseases and disorders including but not limited to arthritis, peripheral artery disease, vasculitis, sepsis, diabetes with end organ damage, cardiovascular disease and CKD
* Currently prescribed immunomodulatory medication or immunocompromised
* Received chemotherapy within 2 weeks of predicted sampling
* Receiving vasopressor support prior to surgery
* History of recent major trauma within the last 2 months (e.g., surgery or injury requiring hospitalisation)

Critically ill patients

* Patients with restricted liberty, prisoners or under legal protection• Anticipated prohibitively difficult venous cannulation
* Presenting with inflammatory diseases and disorders including but not limited to arthritis, peripheral artery disease, vasculitis, diabetes with end organ damage, cardiovascular disease and CKD.
* Currently prescribed immunomodulatory medication or immunocompromised
* Received chemotherapy within 2 weeks of predicted sampling.
* History of recent major trauma within the last 2 months (e.g., surgery or injury requiring hospitalisation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical cohort This cohort will predominantly be made up predominantly of patients undergoing major abdominal surgery (HPB, Gynae Onc and Colorectal) requiring recovery in ICU as part of their cancer treatment.
  Critically unwell cohort This cohort will be made up of emergency admissions to ICU for patients requiring additional organ support.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Differential gene expression in endothelial cells | 2 years
  Using RNA extracted from the two patient cohorts and controls in part 1, we plan to use RNA-SEQ to identify differentially expressed genes. Once we have identified genes we believe to be critically involved with endothelial dysfunction, we will then perform serial sampling on an additional two groups of patients and using qRT-PCR to analyse gene expression changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT06613256/Prot_000.pdf